CLINICAL TRIAL: NCT06308016
Title: Study of the Risk of Pharyngocutaneous Fistula (PCF) in a Population of Patients Undergoing Total Laryngectomy and Creation of a Score for Pre-operative Risk Stratification (Fistula-score)
Brief Title: Study of the Risk of Pharyngocutaneous Fistula in a Population of Patients Undergoing Total Laryngectomy and Creation of a Score for Pre-operative Risk Stratification.
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 25/IRE/23
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Laryngeal Cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter retrospective study of a cohort of patients affected by laryngeal carcinoma and subjected to total laryngectomy surgery at the centers participating in the reference period and responding to inclusion criteria.

DETAILED DESCRIPTION:
Evaluate the relative weight of each factor pre-operative risk, in order to build a score (fistula-score) to be able to stratify before surgery surgical total laryngectomy patients in low-risk and high-risk PCF pharyngocutaneous fistula.

Analyze and process data relating to a total of approximately 500 patients underwent, consecutively, total laryngectomy for malignant neoplasm of the larynx

The results obtained from the present study will allow patients to be stratified into low and high risk for PCF to undergo total laryngectomy, so as to reduce this surgical complication

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing LT surgery with direct closure of the pharynx in case of:

* naïve laryngeal neoplasm (cT1-T3 and cT4a without extension to the esophagus or hypopharynx or oropharynx);
* recurrence of laryngeal neoplasm in a patient who has undergone previous surgical treatment (CO2 laser limited within the larynx or OPHL);
* recurrence of laryngeal neoplasm after RT or Ch-RT treatment;
* lack of functionality of the larynx induced by (Ch-)RT treatment;
* Availability of data according to the assessments that will have to be made, including a FU period of 2 months.

Exclusion Criteria:

* Use of flap, pedicled / free, on-lay / in-lay at the same time as LT surgery. Patients previously subjected to trans-oral surgery of the hypopharynx and/or oropharynx.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the present study, data relating to patients who, in a manner, will be analyzed retrospectively consecutive, I meet the following criteria.
  All patients underwent procedures and/or diagnostic-therapeutic procedures, as well as tests and assessments as required by guidelines and/or conventional clinical management
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Identification of risk factors | 12 months
  The primary objective of the project is the identification of pre-operative risk factors

SECONDARY OUTCOMES:
Stratify patients | 12 months
  The secondary objective is to construct a score to stratify patients according to the risk of developing PCF

CONTACTS AND LOCATIONS:
Overall Officials: Raul Pellini, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy